CLINICAL TRIAL: NCT06768632
Title: Bioequivalence Test of Eltrombopag Olamine Tablets in Humans Under Fasting State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ZDTQ-BE-2019-AQBP
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: single-dose of test formulation+single-dose of reference formulation (Active Comparator): 18 subjects were enrolled, of whom 9received the Investigational drug and 9 received reference preparation.
  Interventions: Drug: Group 1: single-dose of test formulation+single-dose of reference formulation
- Group 2: single-dose of reference formulation+single-dose of test formulation (Active Comparator): 18 subjects were enrolled, of whom 9received the Investigational drug and 9 received reference preparation.
  Interventions: Drug: Group 2: single-dose of reference formulation+single-dose of test formulation

INTERVENTIONS:
Drug: Group 1: single-dose of test formulation+single-dose of reference formulation — Eltrombopag Tablets is a small molecule non peptide thrombopoietin receptor agonist.
  Arms: Group 1: single-dose of test formulation+single-dose of reference formulation
Drug: Group 2: single-dose of reference formulation+single-dose of test formulation — Eltrombopag Tablets is a small molecule non peptide thrombopoietin receptor agonist.
  Arms: Group 2: single-dose of reference formulation+single-dose of test formulation

SUMMARY:
The overall design of this clinical study is a single center, randomized, open label, single dose, two sequence, two cycle bioequivalence trial in healthy individuals under fasting conditions. According to the randomized crossover self-control method, healthy volunteer subjects were orally administered with Eltrombopag Olamine Tablets produced by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. and Reference Listed Drug (RLD) on an empty stomach to evaluate the human bioequivalence of single dose administration, providing reference for their clinical evaluation and medication.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
* Able to complete the study according to the requirements of the trial protocol;
* The participants (including their partners) are willing to voluntarily use effective contraceptive methods within 6 months from screening until the last dose of study drug, as detailed in the Appendix;
* Male and female subjects aged 18-55 years old (including 18 and 55 years old);
* he body weight of male subjects should not be less than 50 kg and the body weight of female subjects should not be less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), BMI in the range of 18-28 kg/m2 (including the cut-off value);
* Health condition: History of no heart, liver, kidney, digestive tract, nervous system, mental disorders, metabolic disorders, etc；
* The physical examination was normal or abnormal without clinical significance.

Exclusion Criteria:

* Smoking more than 5 cigarettes per day in the 3 months before the study;
* Allergic constitution (multi-drug and food allergy);
* A history of drug and/or alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL spirits, or 100 ml wine);
* Donation or massive blood loss (> 400 mL) within 3 months before screening;
* Taking any drugs that alter liver enzyme activity 28 days before screening;
* Have taken any prescription medication, over-the-counter medication, any vitamin product or herbal medicine within 14 days before screening;
* Those who had taken special diet (including dragon fruit, mango, grapefruit, etc.) or had strenuous exercise within 2 weeks before screening, or had other factors affecting drug absorption, distribution, metabolism, and excretion;
* Combined with the following inhibitors or inducers of CYP3A4, P-gp, or Bcrp, such as itraconazole, ketoconazole, or dronedarone;
* A recent major change in diet or exercise habits;
* Have taken a study drug or participated in a clinical trial of the drug within three months before taking the study drug;
* A history of dysphagia or any gastrointestinal disorder affecting drug absorption or a history of cholecystectomy or biliary tract disease;
* Have any condition that increases the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers;
* ECG abnormalities have clinical significance;
* The female subjects were lactating or seropositive for pregnancy during the screening or test period;
* Clinically significant abnormalities on clinical examination or other clinical findings (including but not limited to gastrointestinal, renal, hepatic, neurological, hematologic, endocrine, oncologic, pulmonary, immune, psychiatric, or cardio-cerebrovascular diseases);
* Viral hepatitis (including hepatitis B and C), AIDS antibody, treponema pallidum antibody positive;
* From the screening stage to the onset of acute illness before study medication;
* Consumption of chocolate, any caffeinated or xanthine-rich food or beverage 48 hours before taking the study drug;
* Have taken any alcohol-based product within 24 hours before taking the study medication;
* Individuals who test positive for alcohol and drugs or have a history of drug abuse within the past five years or have used drugs in the three months prior to the experiment;
* Difficulty in blood collection or inability to tolerate venipuncture blood collection;
* The subject is unable or unable to comply with ward management regulations;
* The subject is unable to complete the experiment due to personal reasons;
* Other researchers determine that it is not suitable for selection in this project.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Maximum Concentration
Time to maximum concentration (Tmax) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Time to maximum concentration following drug administration.
Area under the drug-time curve (AUC) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Area under the drug-time curve
Apparent terminal elimination half-life (t1/2) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Apparent terminal elimination half-life following drug administration.
Apparent volume of distribution (Vd/F) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Apparent volume of distribution
Clearance rate (CL/F) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Clearance rate
Apparent terminal elimination rate constant (λz) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Apparent terminal elimination rate constant.
Relative bioavailability (F) | Before administration and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 12, 24, 48, 72 hours after administration
  Relative bioavailability

SECONDARY OUTCOMES:
Incidence of adverse events | From the first dose to the end of follow-up
  Occurrence of all adverse events (AEs), serious adverse events (SAEs), and treatment-related adverse events (TEAEs) were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Lianyungang First People's Hospital, Lianyungang, Jiangsu, China